CLINICAL TRIAL: NCT02329899
Title: Standardisation of Investigations of Mild Bleeding Disorders
Acronym: MBD
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Françoise Boehlen, MD, MD, University Hospital, Geneva
Other Study IDs: 10-246
Record Dates: First submitted 2014-12-22; First posted 2015-01-01 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Hemorrhagic Disorders
MeSH Terms: conditions — Hemorrhagic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 aliquots of plasma from 2x 6 ml EDTA blood 2 aliquots of plasma from 2 x 2.7 ml citrate blood 2 aliquots of plasma from 1 x 4 ml heparin blood Storage at -80°C
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Possible MBD: Defined by:
  * a bleeding score >= 4 in adults;
  * a bleeding score >= 2 in children (for girls, up to menses);
  * a past medical history that include menorrhagia, haemorrhage from the umbilical stump, bleeding at circumcision, cephalhematoma at birth, hematuria, whatever the bleeding score is;
  * a past medical history suggestive of a MBD with no haemostatic challenge and a low bleeding score.
  In this group, the second step of investigations will be performed.
  Interventions: Other: Second step of investigations
- MBD unlikely: Patients without criteria for possible MBD as listed above.
  In this group, no further investigation will be performed if the first step is normal. The second step of investigations will be performed only in case of significant abnormalities in the first step of investigation.
  Interventions: Other: Second step of investigations

INTERVENTIONS:
Other: Second step of investigations — Second step according to results of the first step:
  * exploration of coagulation factors;
  * factor XIII and fibrinolysis investigations;
  * investigation of platelet function;
  * investigation of thrombocytopenia.

SUMMARY:
Observational study aimed at evaluating the clinical impact of a standardised diagnostic procedure for the investigation of patients with suspected mild bleeding disorder (MBD).

DETAILED DESCRIPTION:
The working hypothesis of this prospective diagnostic study is that a standardised procedure in investigating patients with suspected MBD will lead to a better discrimination between patients with and without MBD and a more precise characterisation of MBD.

The primary objective of this diagnostic study is to evaluate the efficiency of a standardised procedure of MBD in children and adults referred to their respective outpatient clinics for bleeding symptoms. The following endpoints will be evaluated:

1. The relative number of precise diagnosis (according to recognised classification of haemostatic disorders) in each clinical probability category;
2. The number of biological tests performed per patient in each clinical probability category;
3. The relative number of patients with no specialised investigations in the low risk group.

The secondary objective is to evaluate the bleeding events during a one-year follow-up. Follow-up will be performed with a phone call one year after the last consultation of the patient. The definition of a bleeding event will be any bleeding that promotes any specific medical attention (consultation, hospitalisation, transfusion, re-intervention in case of surgery). The detailed clinical history regarding each event will be collected. Bleeding events will be correlated to the clinical probability assessed at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged more than two years-old referred by their physician (gynaecologist, paediatrician, general practitioner, surgeon, etc.) for investigations of a possible bleeding tendency will be included in this study. This prospective study will include consecutive patients attending the four outpatient clinics (Division of Angiology and Haemostasis and Paediatric Onco-Haematology Unit, University Hospitals of Geneva).

Exclusion Criteria:

* Pregnant women will be excluded because of modifications of the known modifications of the haemostasis system during pregnancy. Adult patients without discernment capacity will be excluded.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (children or adults) referred to a tertiary care center (haemostasis unit) for investigation of mild bleeding symptoms (with suspicion of mild bleeding disorder)
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2012-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Relative number of precise diagnosis | after the completion of the standardized diagnostic procedure (on average 6 weeks after enrollment)
  Diagnosis are going to be evaluated according to recognized classification of haemostatic disorders
Number of biological tests performed per patient | after the completion of the standardized diagnostic procedure (on average 6 weeks after enrollment)
Relative number of patients with no specialised investigations in the low risk group | after the completion of the standardized diagnostic procedure (on average 1 week after enrollment in this low risk group)

SECONDARY OUTCOMES:
Evaluation of bleeding events | After one year follow-up
  Phone call

CONTACTS AND LOCATIONS:
Overall Officials: Boehlen Francoise, MD, Principal Investigator — Haemostasis unit, University Hospitals of Geneva, Switerland
Locations (1):
- Haemostasis unit, University Hospitals of Geneva, Geneva, Switzerland